CLINICAL TRIAL: NCT05458362
Title: Efficacy of the Mobile App Augmentation to a Brief Anxiety Sensitivity Treatment
Brief Title: Brief Enhanced Anxiety Sensitivity Treatment (Group)
Acronym: Group BEAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, Nicholas Allan, Assistant Professor of Clinical Psychology, Ohio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Group_BEAST
Record Dates: First submitted 2022-05-06; First posted 2022-07-14 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Anxiety Sensitivity; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A 1.5-hour intervention session will be completed by all participants. We will ask all participants to complete homework exposure exercises. They will receive phone app reminders about completing homework.
  Treatment group (EMI group): For two weeks after the session, four times a day, the EMI group will receive prompts via the HIPAA-compliant EMI application (metricwire.com). The prompts will ask them about their current anxiety level. If they endorse elevated anxiety, they will be provided with a brief message reminding them about the coping skills covered during the session. They will also receive daily prompts to do exposures and enter the results in the app.
  Control group: The control group will not receive EMI prompts and will be offered to complete EMI after the follow-up assessment.
Masking Description: During the consent process, participants are provided information that some of them may receive additional phone app intervention. This is not stressed at any other time during the study. After randomization has been completed, treatment session groups will be formed including participants from both conditions. After the the session, participants receive an email reminding them about the surveys and reminders they will be getting through the app during the upcoming 2 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMI group (Experimental): For two weeks after the intervention session, participants will report on their anxiety level four times per day. When participants endorse elevated anxiety, they will receive a message relevant to their most stressful symptom at the moment reminding them of the topics covered in the intervention session.
  As the efficacy of the EMI component is being tested, only the EMI group will receive EMI.
  Interventions: Behavioral: Brief Enhanced Anxiety Sensitivity Treatment (Group BEAST)
- Control group (Active Comparator): The control group will not receive EMI prompts and will be offered to complete EMI after the follow-up assessment.
  Interventions: Behavioral: Control group Anxiety Sensitivity Treatment

INTERVENTIONS:
Behavioral: Brief Enhanced Anxiety Sensitivity Treatment (Group BEAST) — Group BEAST consists of a 1.5-hour-long intervention session, followed by a 2-week-long EMI. During the intervention session, participants will receive psychoeducation (e.g., defining common terms like anxiety and stress), discuss popular misconceptions they may have about anxiety symptoms, and complete exposure exercises (e.g., practicing facing feared physical sensations such as trembling or elevated heart rate). Homework exposure exercises will be completed by all participants. They will receive phone app reminders about completing homework.
  Only the EMI group will receive EMI prompts and intervention.
  Arms: EMI group
Behavioral: Control group Anxiety Sensitivity Treatment — Control group Anxiety Sensitivity Treatment consists of a 1.5-hour-long intervention session, followed by a 2-week-long EMI. During the intervention session, participants will receive psychoeducation (e.g., defining common terms like anxiety and stress), discuss popular misconceptions they may have about anxiety symptoms, and complete exposure exercises (e.g., practicing facing feared physical sensations such as trembling or elevated heart rate). Homework exposure exercises will be completed by all participants. They will receive phone app reminders about completing homework.
  Arms: Control group

SUMMARY:
One-third of the U.S. population experience anxiety disorders in their lifetime and only 25% of them seek treatment, reporting logistics and cost of treatment among the primary barriers. A potential way to prevent and treat multiple anxiety disorders is to target the risk factors that contribute to their etiology. One such well-researched risk factor is anxiety sensitivity (AS), a fear of anxiety-related sensations. Given a need for affordable and accessible brief treatments, we and our colleagues have been iteratively developing Brief Enhanced Anxiety Sensitivity Treatment (BEAST), a one-session virtual treatment targeting AS. Older versions of BEAST include psychoeducation, interoceptive exposure (IE), and IE homework. Several studies showed that the previous versions of BEAST reduced AS and, through the reductions in AS, they also reduced anxiety. However, the effect sizes for the decrease in anxiety were modest. Efficacy and personalization may be improved using Ecological Momentary Intervention (EMI). EMI delivers brief interventions remotely in real-time and in natural settings. The goal of the current study is to test the efficacy of adding EMI to BEAST. Participants will be randomly assigned to EMI and control (no EMI) conditions. All participants will receive a virtual 1.5-hour-long intervention group session facilitated by a therapist. The EMI group will receive individualized intervention messages helping them to use new skills for two weeks after the session. After the two-week EMI period, all participants will complete post-treatment measures of AS and anxiety. A month later, they will complete a follow-up assessing AS and anxiety. The efficacy of the EMI component in reducing AS and anxiety will be tested using multilevel modeling. Improving the efficacy of BEAST, while keeping it brief, affordable, and accessible online, is an important step towards making it a treatment that may be used on a large scale.

DETAILED DESCRIPTION:
There is a high need for prevention and treatment of anxiety disorders and for more accessible and affordable treatments. Targeting a risk factor for development and maintenance of multiple anxiety disorders may be an efficient way to prevent and treat anxiety. Anxiety sensitivity (AS)-the fear of anxiety sensations because of the belief that these sensations may lead to catastrophic outcomes-is a potent prevention and treatment target because it predicts development and maintenance of anxiety over time. Anxiety Sensitivity Amelioration Training (ASAT) is an ultra-brief, affordable treatment delivered virtually that targets AS. ASAT is a potent prevention and treatment protocol that reduces anxiety by reducing AS. However, the effect sizes were modest.

Adding Ecological Momentary Intervention (EMI) to the treatment could motivate the participants to apply skills they learned in treatment in a variety of real-life situations and to practice homework exercises. EMI delivers the intervention remotely in real-time and in natural settings, providing better learning through deeper processing. EMI alone is an effective treatment for anxiety and has been an efficacious enhancement to a 6-session treatment for generalized anxiety disorder. However, adding EMI to a 6-session panic disorder treatment did not improve the efficacy of the intervention. Because EMI can reduce anxiety as a stand-alone treatment and due to the inconclusive results about the efficacy of EMI as an added component, it is important to test the effect of adding EMI to the ASAT. We called the treatment including EMI the Brief Enhanced Anxiety Sensitivity Treatment (BEAST).

The goal of this study is to compare the efficacy of the BEAST with and without the EMI component. Interventions will be delivered to the adult community members and students in Athens, Ohio. Based on the power analysis, 75 adult participants will be recruited using email and online advertising. Based on methods used in the prior studies and the current design, inclusion criteria are elevated AS symptoms, access to a smartphone with internet connection. Exclusion criteria are heart disease, respiratory disorders, renal disease, seizure disorder, uncontrolled hypertension or migraines, current substance use disorder (severe), uncontrolled manic or psychotic symptoms, and suicidal ideation that requires hospitalization. All participants will receive a one-hour manualized group intervention educating about anxiety as an alarm system, the benign nature of anxiety sensations, myth-busting, and modifying biases about feared stimuli. The session will also include therapist-guided interoceptive exposure. Participants will be asked to do the exposure at home at least once a day for two weeks. For two weeks after the session, four times a day, the EMI group will receive prompts via the HIPAA-compliant EMI application (metricwire.com). The prompts will ask them about their current anxiety level. If they endorse elevated anxiety, they will be provided with a brief message reminding them about the coping skills covered during the session. They will also receive daily prompts to do exposures and enter the results in the app. The control group will not receive the EMI prompts and will be offered to complete EMI four weeks after the treatment. The intervention will be delivered by graduate students in a clinical Ph.D. program using Microsoft Teams, in groups of 4-6 participants.

AS and anxiety will be assessed using online questionnaires at baseline, at week two and week six after the delivery of the intervention session. Brief interview will be administered at baseline to assess the pathology listed in the exclusion criteria. Multilevel modeling will be used compare AS and anxiety between the groups at both follow-ups controlling for the baseline AS and anxiety. BEAST is an affordable intervention that can be used for prevention and treatment of anxiety and can be administered virtually. This is the first study testing the efficacy an added EMI component to a one-session-long anxiety intervention.

ELIGIBILITY:
Inclusion Criteria:

* elevated anxiety sensitivity symptoms (i.e., ASI-3 scores greater than or equal to 17),
* have access to a device smartphone with internet connection.

Exclusion Criteria:

* cardiovascular disease or stroke
* respiratory disorders (asthma, COPD, other),
* renal disease,
* epilepsy or other seizure disorder,
* and uncontrolled hypertension or migraines.
* current substance use disorder (severe),
* uncontrolled manic symptoms,
* uncontrolled psychotic symptoms,
* suicidal ideation that requires hospitalization,
* if the participants endorse that English is not their first language in the screening questionnaire and demonstrate significant impairment in understanding the interviewer, they will be considered not proficient in English and will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety Sensitivity Inventory-3 (ASI-3; Taylor et al., 2007) | Screening, baseline, post-treatment including EMI (2 weeks after the session), 1 month follow-up.
  The ASI-3 is an 18-item self-report questionnaire of anxiety sensitivity measured on a 5-point Likert-like scale ranging from 0 (very little) to 4 (very much).
Change in PROMIS Anxiety scale - 8a | Baseline, post-treatment including EMI (2 weeks after the session), 1 month follow-up.
  The PROMIS Anxiety scale measures anxiety broadly, including items to assess fear, anxious misery, hyperarousal, and somatic symptoms. Items are on a 5-point scale from 1 (Never) to 5 (Always).

SECONDARY OUTCOMES:
Change multiple times a day - EMI anxiety questions (EMI group) | 2 weeks of EMI - 4 times a day
  On every EMI measurement occasion, participants will be asked to report their level of anxiety using the question "How anxious are you?" on a scale ranging from 0 to 100. If they endorse elevated anxiety of 30 or above (Newman et al., 2014), they will be sent another question: What stressful symptoms are you experiencing? (a) Body sensations, (b) Mind and concentration, (c) Concerned about being judged for your anxiety symptoms. Next, they will be asked to choose a specific symptom from the dimension they have picked. Based on this symptom, they will be shown a message offering a CBT strategy to cope with the symptom and the distress effectively.
  We will be sending the prompt 80% of the time when an elevated symptom level is reported (30-100 on a sliding scale) and provide intervention in 10% of cases when a low level of the symptom is reported (0-29 on a sliding scale).
Daily change - Short Scale Anxiety Sensitivity Index (all participants) | 2 weeks of EMI - 1 time a day
  SSASI is a short version of the ASI-3 (Taylor et al., 2007). It is a 5-item questionnaire measuring AS on a 5-item Likert scale from 0 (very little) to 4 (very much). The SSASI has items corresponding to all three dimensions of AS: Physical concerns, cognitive concerns, and social concerns. This measure will be added to the first EMI prompt of the day. This will allow us to measure the change in the participants AS symptoms daily. The SSASI will be modified to assess symptoms during the past 24 hours.
Daily change - PROMIS Anxiety Short Form 8a Modified (all participants) | 2 weeks of EMI - 1 time a day
  The PROMIS Anxiety Short Form will be modified to assess anxiety symptoms the participant has experienced yesterday as opposed to 7 past days. This measure will be added to the first EMI prompt of the day. This will allow us to measure the change in the participants anxiety symptoms daily.

OTHER OUTCOMES:
Demographic questionnaire | Baseline
  The demographic questionnaire will include questions about age, sex at birth, gender, sexual orientation, race, ethnicity, marital status, number of children, education, employment status, occupation, income, and rural/urban geographic area. Participants will be asked if they have contracted COVID-19 and how severe their symptoms were.
Change in PROMIS Depression scale - 8a | Baseline, post-treatment including EMI (2 weeks after the session), 1 month follow-up.
  The PROMIS Depression scale is an 8-item measure of depression. Items are on a 5-point scale from 1 (Never) to 5 (Always).
Change in PROMIS Psychological Stress scale - 8a | Baseline, post-treatment including EMI (2 weeks after the session), 1 month follow-up.
  The PROMIS Psychological Stress scale is an 8-item tool assessing feelings about self and the world in the context of challenges. Items are on a 5-point scale from 1 (Never) to 5 (Always).
COVID-19 impact battery short-form | Baseline
  COVID-19 impact battery short-form (CIB-SF baseline only): A five item questionnaire designed by the investigators will be used to assess COVID-19 related worries and impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allan NP, Capron DW, Lejuez CW, Reynolds EK, MacPherson L, Schmidt NB. Developmental trajectories of anxiety symptoms in early adolescence: the influence of anxiety sensitivity. J Abnorm Child Psychol. 2014 May;42(4):589-600. doi: 10.1007/s10802-013-9806-0. PMID 24062146
- [Background] Goetter EM, Frumkin MR, Palitz SA, Swee MB, Baker AW, Bui E, Simon NM. Barriers to mental health treatment among individuals with social anxiety disorder and generalized anxiety disorder. Psychol Serv. 2020 Feb;17(1):5-12. doi: 10.1037/ser0000254. Epub 2018 Aug 2. PMID 30070552
- [Background] Heron KE, Smyth JM. Ecological momentary interventions: incorporating mobile technology into psychosocial and health behaviour treatments. Br J Health Psychol. 2010 Feb;15(Pt 1):1-39. doi: 10.1348/135910709X466063. Epub 2009 Jul 28. PMID 19646331
- [Background] Kenardy JA, Dow MG, Johnston DW, Newman MG, Thomson A, Taylor CB. A comparison of delivery methods of cognitive-behavioral therapy for panic disorder: an international multicenter trial. J Consult Clin Psychol. 2003 Dec;71(6):1068-75. doi: 10.1037/0022-006X.71.6.1068. PMID 14622082
- [Background] Keough ME, Schmidt NB. Refinement of a brief anxiety sensitivity reduction intervention. J Consult Clin Psychol. 2012 Oct;80(5):766-72. doi: 10.1037/a0027961. Epub 2012 Apr 2. PMID 22468909
- [Background] Kessler RC, Aguilar-Gaxiola S, Alonso J, Chatterji S, Lee S, Ormel J, Ustun TB, Wang PS. The global burden of mental disorders: an update from the WHO World Mental Health (WMH) surveys. Epidemiol Psichiatr Soc. 2009 Jan-Mar;18(1):23-33. doi: 10.1017/s1121189x00001421. PMID 19378696
- [Background] Kessler RC, Petukhova M, Sampson NA, Zaslavsky AM, Wittchen H -U. Twelve-month and lifetime prevalence and lifetime morbid risk of anxiety and mood disorders in the United States. Int J Methods Psychiatr Res. 2012 Sep;21(3):169-84. doi: 10.1002/mpr.1359. Epub 2012 Aug 1. PMID 22865617
- [Background] LaFreniere LS, Newman MG. A BRIEF ECOLOGICAL MOMENTARY INTERVENTION FOR GENERALIZED ANXIETY DISORDER: A RANDOMIZED CONTROLLED TRIAL OF THE WORRY OUTCOME JOURNAL. Depress Anxiety. 2016 Sep;33(9):829-39. doi: 10.1002/da.22507. Epub 2016 Apr 7. PMID 27062682
- [Background] Newman MG, Przeworski A, Consoli AJ, Taylor CB. A randomized controlled trial of ecological momentary intervention plus brief group therapy for generalized anxiety disorder. Psychotherapy (Chic). 2014 Jun;51(2):198-206. doi: 10.1037/a0032519. Epub 2013 Sep 23. PMID 24059730
- [Background] Schmidt NB, Capron DW, Raines AM, Allan NP. Randomized clinical trial evaluating the efficacy of a brief intervention targeting anxiety sensitivity cognitive concerns. J Consult Clin Psychol. 2014 Dec;82(6):1023-33. doi: 10.1037/a0036651. Epub 2014 May 12. PMID 24821096
- [Background] Schmidt NB, Eggleston AM, Woolaway-Bickel K, Fitzpatrick KK, Vasey MW, Richey JA. Anxiety Sensitivity Amelioration Training (ASAT): a longitudinal primary prevention program targeting cognitive vulnerability. J Anxiety Disord. 2007;21(3):302-19. doi: 10.1016/j.janxdis.2006.06.002. Epub 2006 Aug 4. PMID 16889931
- [Background] Schmidt NB, Mitchell MA, Richey JA. Anxiety sensitivity as an incremental predictor of later anxiety symptoms and syndromes. Compr Psychiatry. 2008 Jul-Aug;49(4):407-12. doi: 10.1016/j.comppsych.2007.12.004. Epub 2008 Mar 19. PMID 18555063
- [Background] Wang PS, Lane M, Olfson M, Pincus HA, Wells KB, Kessler RC. Twelve-month use of mental health services in the United States: results from the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):629-40. doi: 10.1001/archpsyc.62.6.629. PMID 15939840